CLINICAL TRIAL: NCT07121842
Title: GLIMPCE: Glioblastoma Imaging for the Detection of Tumor Progression Using APTw-CEST MRI
Brief Title: Glioblastoma Imaging for the Detection of Tumor Progression Using APTw-CEST MRI
Acronym: GLIMPCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: UMC Utrecht (Other); LeidenUMC (Unknown); Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Esther Warnert, Assistant Professor, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL86895.078.24
Record Dates: First submitted 2025-07-31; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; MRI; CEST; Pseudoprogression; multi-center; APTw-CEST
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Extended MRI (Other): The MRI protocol for every clinical MRI scan taken in follow-up is extended with 15 minutes.
  Interventions: Diagnostic Test: Extended MRI

INTERVENTIONS:
Diagnostic Test: Extended MRI — The MRI protocol for every clinical follow-up MRI scan is extended with 15 minutes to add the APTw-CEST scan.

SUMMARY:
In this study, the invesigators look at how a new MRI technique (called amide proton transfer weighted (APTw) chemical exchange saturation transfer (CEST)) can improve treatment for brain tumors through early detection of tumor progression after radiotherapy and/or chemotherapy treatment.

An issue with the current treatment for patients with a brain tumor, is the inability to detect tumor progression early. An abnormality is seen on MRI scans taken shortly after treatment with radiotherapy in about 30% of patients.

This abnormality may be a sign that radiotherapy treatment has worked well and will disappear on its own after a while. However, an abnormality can also be a sign of active tumor tissue. Then it shows that the treatment has not worked well enough. When there is active tumor tissue, this is called 'tumor progression'. When there is an abnormality that disappears on its own after a while, there is no active tumor tissue. This is called 'pseudoprogression'.

Currently, there are two options to determine whether tumor progression or pseudoprogression has taken place: Do another brain surgery to see if the abnormality contains active tumor tissue or wait and have regular MRI scans until it is clear whether the abnormality goes away on its own.

Amide proton transfer weighted chemical exchange saturation transfer (APTw-CEST) imaging is a new MRI technique in which investigators can produce images that show the accumulation of protein. APTw-CEST has previously been shown to be able to distinguish tumor progression from pseudoprogression earlier than current standard MRI scans. However, these previous studies have drawbacks: they were either done with a small group of patients in 1 hospital, or with a 7 Tesla MRI scanner, a rare type of scanner not standard in hospitals, or done in animal models.

In this research project the investigators now want to prepare APTw-CEST for standard patient care for patients with glioblastoma in the Netherlands so that in the future APTw-CEST can be included as a standard scan during treatment. The investigators are doing this by introducing APTw-CEST MRI on the clinical MRI scanners of four different hospitals. Ultimately, the investigators want to use this to create national guidelines for measuring and viewing APTw-CEST MRI images for early detection of tumor progression.

DETAILED DESCRIPTION:
Rationale:

A major issue with glioblastoma treatment is the occurrence of contrast enhancement after treatment with radiotherapy or chemoradiotherapy. This enhancement can be due to more tumor growth; called true progression. It can also be due to treatment-related effects; called pseudoprogression. Amide proton transfer weighted (APTw) chemical exchange saturation transfer (CEST) magnetic resonance imaging (MRI) is a technique that indirectly images proteins and peptides in a tissue. Because these molecules are overexpressed in tumor tissue, APTw-CEST MRI has been shown to be good at distinguishing between true progression and pseudoprogression, which is important as they require vastly different responses. This technique shows promise to become an important biomarker in glioblastoma treatment, how-ever it currently lacks standardization, as studies are generally done in one center on MRI machines of one vendor.

This multi-center study will make APTw-CEST MRI a clinically usable biomarker for the detection of tumor progression in glioblastoma patients by providing acquisition and post-processing recommendations, as well as a threshold on APTw-CEST images that would allow a clinician to accurately distinguish between pseudoprogression and true progression, regard-less of where the images were acquired and with which system.

The underlying processes that make APTw-CEST a reliable biomarker for glioblastoma treatment response evaluation are not clearly known. Using other advanced MRI techniques (diffusion, perfusion) and O-(2-[18F]fluoroethyl-)-L-tyrosine Positron Emission Tomography (FET-PET), and correlating these images with the APTw-CEST images will give a better insight into these processes.

Primary Objective: Determine the optimal threshold on APTw-CEST images in a multi-center (4 academic institutes) multi-vendor (Philips, Siemens and GE) clinical trial, to distinguish tumor progression from treatment-related effects.

Secondary Objective(s):

* Correlate APTw-CEST MRI to complimentary, advanced imaging parameters such as FET-PET, diffusion and perfusion MRI, and Response Assessment for Neuro-Oncology (RANO) criteria.
* Provide recommendations for the acquisition and post-processing of APTw-CEST MRI.

Study design:

In this prospective cohort study, all clinical MRI scans will be extended with the APTw-CEST protocol. The patient receives their standard care and decisions will be made based on standard-of-care imaging. The APTw-CEST images and diagnosis from standard follow-up will be used to determine the threshold on APTw-CEST images that would most accurately distinguish between pseudoprogression and true progression early after treatment.

Additional advanced imaging (diffusion, perfusion, FET-PET) taken during the treatment and follow-up of the patient will be used to correlate areas of high APTw signal with other signals.

Study population: 120 patients diagnosed with or suspected of glioblastoma using molecular or histochemistry analysis or medical imaging respectively.

Intervention (if applicable): Each patient will have extensions to all MRI scans taken for the treatment and follow-up of glioblastoma. The APTw-CEST sequence will be added to all clinical scans, for an addition of 10-15 minutes of scan time.

Main study parameters/endpoints: Threshold on APTw-CEST images that accurately distinguishes between true progression and pseudoprogression in recently treated glioblastoma patients. The accuracy will be optimized using Receiver operating characteristic (ROC) curve analysis and the Youden index.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The clinical care of the patient group will not be altered. The APTw-CEST images will not be used to make any clinical decision. Patients will not have personal benefit from this study, and will have the burden of a prolonged scan time of 10-15 minutes. All further imaging used in this study; perfusion, diffusion and FET-PET will not be taken specifically for this study and will only be taken when clinically indicated, except in LUMC where the FET-PET will be added to standard-of-care. The addition of FET-PET in the patient group in LUMC is warranted as the long-term risks are negligible for this patient group, due to the median survival of 12-14 months.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of glioblastoma based on histopathological or molecular analysis of biopsy after surgery, or suspected of glioblastoma based on medical imaging.
* Scheduled to undergo radiotherapy or combined chemo-and radiotherapy
* 18 years and older
* Able to give informed consent.
* Patient will undergo clinically indicated MRIs

Exclusion Criteria:

* Not able to give informed consent
* Contraindication for MRI
* Brain pathology affecting CEST contrast, such as recent stroke or earlier cranial radiotherapy, as determined by the principal investigators (PIs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Determining the Threshold | Until 1 year after the first MRI scan with the additional APTw-CEST added
  Determine the optimal threshold on APTw-CEST images in a multi-center (4 aca-demic institutes) multi-vendor (Philips, Siemens and GE) clinical trial, to distinguish tumor progression from treatment-related effects.

SECONDARY OUTCOMES:
Correlations with other MRI and PET scans. | Up until 1 year from the date of the first MRI scan with added APTw-CEST
  Correlate APTw-CEST MRI to complimentary, advanced imaging parameters such as FET-PET, diffusion and perfusion MRI, and RANO criteria.

CONTACTS AND LOCATIONS:
Locations (4):
- Netherlands (4):
  - Amsterdam UMC, Amsterdam
  - Leiden UMC, Leiden
  - Erasmus MC, Rotterdam
  - UMC Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://iknl.nl/kankersoorten/hersentumoren/registratie/incidentie
- See also: Related Info — https://iknl.nl/nieuws/2019/glioomzorg-in-nederland